CLINICAL TRIAL: NCT01509547
Title: A Randomized Controlled Trial of Varenicline for Adolescent Smoking Cessation
Brief Title: Varenicline for Adolescent Smoking Cessation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Kevin Gray, MD, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00014398
Record Dates: First submitted 2011-12-14; First posted 2012-01-13 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- varenicline (Experimental): Participants >55 kg will take varenicline 0.5 mg once daily for 3 days, titrated to 0.5 mg twice daily for 4 days, titrated to 1 mg twice daily for 11 weeks. Participants ≤55 kg will take varenicline 0.5 mg once daily for 7 days, titrated to 0.5 mg twice daily for 11 weeks.
  Interventions: Drug: Varenicline
- placebo (Placebo Comparator): Participants >55 kg will take placebo 0.5 mg once daily for 3 days, titrated to 0.5 mg twice daily for 4 days, titrated to 1 mg twice daily for 11 weeks. Participants ≤55 kg will take placebo 0.5 mg once daily for 7 days, titrated to 0.5 mg twice daily for 11 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Varenicline — participants >55 kg will take varenicline/placebo 0.5 mg once daily for 3 days, titrated to 0.5 mg twice daily for 4 days, titrated to 1 mg twice daily thereafter. Participants ≤55 kg will take varenicline/placebo 0.5 mg once daily for 7 days, titrated to 0.5 mg twice daily thereafter.
  Other Names: Chantix
  Arms: varenicline
Drug: placebo — participants >55 kg will take varenicline/placebo 0.5 mg once daily for 3 days, titrated to 0.5 mg twice daily for 4 days, titrated to 1 mg twice daily thereafter. Participants ≤55 kg will take varenicline/placebo 0.5 mg once daily for 7 days, titrated to 0.5 mg twice daily thereafter.
  Arms: placebo

SUMMARY:
This is a placebo-controlled smoking cessation treatment study for adolescents ages 14-21. After assessment and inclusion into the study, participants will be randomized to receive a 12-week double blind course of varenicline or placebo.

DETAILED DESCRIPTION:
The objective of this protocol is to examine the efficacy and safety of varenicline for smoking cessation in adolescents. The guiding design philosophy was to model the adult smoking cessation literature (allowing for indirect comparisons of efficacy in different populations) while fine-tuning some elements specifically geared for adolescents. After assessment and inclusion into the study, participants will be randomized to receive a 12-week double blind course of varenicline or placebo. Participants will provide smoking self-report (cigarettes per day) throughout the study. Biological confirmation with carbon monoxide breathalyzer will occur at all visits, and urine cotinine measurement will occur at key time points (baseline, end of treatment and final post-treatment follow-up). Psychiatric/medical visits will occur weekly throughout active treatment to systematically monitor safety and tolerability. After the 12-week treatment course, participants will return for 3 post-treatment follow-up visits (Week 13, Week 18, and Week 26).

ELIGIBILITY:
Inclusion Criteria:

* Age 14-21
* Daily smoker for ≥6 months
* Desire to quit smoking, with at least one prior failed quit attempt and willingness to participate in a treatment study
* If under age 18, parent(s) or guardian(s) able to participate in informed consent and initial assessment (unless the participant provides evidence of emancipated status)
* If female, agreement to use birth control (any form of hormonal contraception such as Depo-Provera, daily oral contraception, transdermal patch, or Nuva-ring; intrauterine device; sterilization; or double barrier contraception, which is a combination of any two of the following methods: condoms, spermicide, diaphragm) to avoid pregnancy

Exclusion Criteria:

* Lifetime history of any DSM-IV-TR mood or psychotic disorder (e.g., major depressive disorder, bipolar disorder, schizophrenia)
* Lifetime history of suicidality, homicidality, or clinically significant hostility/aggression
* Current substance dependence, other than nicotine
* Current unstable major medical disorder
* Current pregnancy or breastfeeding
* Current use of medications with smoking cessation efficacy
* Known hypersensitivity to varenicline

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 157 (Actual)
Dates: Start 2012-08; Primary Completion 2018-01-26 (Actual); Study Completion 2018-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Gray, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902
- [Derived] Gray KM, Baker NL, McClure EA, Tomko RL, Squeglia LM, Saladin ME, Carpenter MJ. Efficacy and Safety of Varenicline for Adolescent Smoking Cessation: A Randomized Clinical Trial. JAMA Pediatr. 2019 Dec 1;173(12):1146-1153. doi: 10.1001/jamapediatrics.2019.3553. PMID 31609433

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 77 | 80
Completed | 42 | 41
Not Completed | 35 | 39
Not completed — Lost to Follow-up | 24 | 14
Not completed — Withdrawal by Subject | 11 | 24
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 77 | 80 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.1 (1.5) | 19.1 (1.4) | 19.1 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 35 | 63
  Male | 49 | 45 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 74 | 79 | 153
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 11 | 22
  White | 54 | 66 | 120
  More than one race | 8 | 3 | 11
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 77 | 80 | 157

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cotinine-confirmed 7-day Point Prevalence Abstinence at the End of Treatment
Description: Self-reported 7-day cigarette abstinence, confirmed by urine corinne ≤50 ng/mL at the end-of-treatment (week 12) visit
Time Frame: 7 days at end of treatment
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 77 | 80
Participants | 4 | 4

2. Primary Outcome: Number of Participants Experiencing Treatment-emergent Adverse Events
Description: Clinician-collected adverse events (regardless of relatedness to medication) occurring at any point after randomization and initiation of treatment.
Time Frame: 26 weeks (12 weeks of treatment plus full post-treatment follow-up)
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 77 | 80
Participants | 55 | 60

3. Secondary Outcome: Percentage of Visits With Abstinence During Treatment
Description: Self-reported between-visit abstinence at weekly visits during treatment (reported as percentage of total possible visits across all participants at which participants self-reported abstinence). Missing data were imputed to non-abstinence.
Time Frame: 12 weeks (all of active treatment)
Measure: Number (95% Confidence Interval); unit: percentage of visits with abstinence
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 77 | 80
percentage of visits with abstinence | 14.2 [11.9 to 16.4] | 7.3 [5.6 to 8.9]

4. Secondary Outcome: Percentage of Post-treatment Visits With Abstinence
Description: Self-reported abstinence at post-treatment follow-up visits (reported as percentage of total possible post-treatment follow-up visits at which abstinence in the prior week was self-reported). Missing data were imputed to non-abstinence.
Time Frame: One week abstinence at the Week 16 and Week 26 post-treatment follow-up visits
Measure: Number (95% Confidence Interval); unit: percentage of visits with abstinence
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 77 | 80
percentage of visits with abstinence | 20.8 [14.4 to 27.2] | 10.6 [5.8 to 15.4]

5. Secondary Outcome: Number of Participants Achieving 7+ Days Abstinence at Any Point During Treatment
Description: Number of participants achieving 7+ days of self-reported abstinence at any point during active treatment
Time Frame: 12 weeks of active treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 77 | 80
Participants | 31 | 24

ADVERSE EVENTS:
Time Frame: 6 months (randomization to last post-treatment follow-up visit)
Description: Assessed and coded in MedDRA terminology by the medical clinician at each visit.
Arm/Group | Varenicline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/80
Other Adverse Events (participants affected / at risk) | 55/77 | 60/80
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=77) | Placebo (N=80)
ear congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1)
blurred vision (Eye disorders) | 1 (1) | 0 (0)
conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
dyspepsia (worsening) (Gastrointestinal disorders) | 2 (2) | 1 (1)
flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
GERD (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastroenteritis (Gastrointestinal disorders) | 1 (1) | 3 (3)
nausea (Gastrointestinal disorders) | 24 (28) | 15 (15)
salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1)
stomachache (Gastrointestinal disorders) | 3 (3) | 0 (0)
stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 11 (15) | 6 (7)
fatigue (General disorders) | 1 (1) | 3 (3)
chest pain (General disorders) | 1 (1) | 1 (1)
boil (Infections and infestations) | 3 (5) | 0 (0)
bronchitis (Infections and infestations) | 4 (4) | 2 (2)
cellulitis (Infections and infestations) | 1 (1) | 1 (1)
folliculitis (Infections and infestations) | 0 (0) | 1 (1)
gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
influenza (Infections and infestations) | 2 (2) | 0 (0)
influenza like illness (Infections and infestations) | 1 (1) | 2 (2)
laryngitis (Infections and infestations) | 0 (0) | 1 (1)
lung infection (Infections and infestations) | 0 (0) | 1 (1)
oral herpes (Infections and infestations) | 0 (0) | 1 (1)
otitis media (Infections and infestations) | 0 (0) | 1 (1)
pharyngitis (Infections and infestations) | 2 (2) | 4 (4)
pneumonia (Infections and infestations) | 1 (1) | 0 (0)
sinusitis (Infections and infestations) | 4 (4) | 1 (1)
urinary tract infection (Infections and infestations) | 0 (0) | 1 (2)
vaginal infection (Infections and infestations) | 0 (0) | 3 (3)
viral upper respiratory tract infection (Infections and infestations) | 21 (25) | 13 (15)
contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
fractured coccyx (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
pain in extremity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
post operative pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
post procedural complication (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
sprained ankle (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
increased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
back muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
foot pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
knee pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
convulsion (Nervous system disorders) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 1 (1)
dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
headache (Nervous system disorders) | 8 (8) | 9 (13)
lightheadedness (Nervous system disorders) | 1 (3) | 1 (2)
memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
migraine (Nervous system disorders) | 0 (0) | 1 (2)
migraine (worsening) (Nervous system disorders) | 0 (0) | 1 (1)
paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
poor quality sleep (Nervous system disorders) | 3 (3) | 0 (0)
somnolence (Nervous system disorders) | 0 (0) | 1 (1)
agitation (Psychiatric disorders) | 8 (9) | 5 (6)
anxiety (Psychiatric disorders) | 1 (1) | 3 (3)
anxiety (worsening) (Psychiatric disorders) | 1 (1) | 1 (1)
attention-deficit/hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0)
depressed mood (Psychiatric disorders) | 3 (3) | 5 (5)
hostility (Psychiatric disorders) | 1 (1) | 1 (1)
hypervigilance (Psychiatric disorders) | 1 (1) | 0 (0)
inappropriate affect (Psychiatric disorders) | 1 (1) | 0 (0)
insomnia (Psychiatric disorders) | 9 (10) | 7 (7)
irritability (Psychiatric disorders) | 0 (0) | 1 (1)
mood swings (Psychiatric disorders) | 1 (1) | 2 (2)
panic attack (worsening) (Psychiatric disorders) | 1 (2) | 0 (0)
passive suicidal ideation (Psychiatric disorders) | 1 (1) | 3 (3)
tobacco withdrawal symptoms (Psychiatric disorders) | 1 (1) | 0 (0)
vivid dreams (Psychiatric disorders) | 10 (10) | 7 (7)
dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 1 (1)
menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
chest congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8)
lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 4 (4)
rhinitis seasonal (worsening) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5)
throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
rash generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT01509547/Prot_SAP_000.pdf
  • Informed Consent Form (2016-06-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT01509547/ICF_001.pdf